CLINICAL TRIAL: NCT01609127
Title: A Randomized, Phase II Study of Tesetaxel Once Every 3 Weeks Versus Tesetaxel Once Weekly for 3 Weeks Versus Capecitabine Twice Daily for 14 Days as First-line Therapy for Subjects With Locally Advanced or Metastatic Breast Cancer
Brief Title: Tesetaxel Every 3 Weeks vs Weekly vs Capecitabine as 1st-line Therapy for Locally Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOB206
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Locally Advanced Non-resectable Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tesetaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tesetaxel every 3 weeks (Experimental): Tesetaxel 27 mg/m2 orally on Day 1 in a 21-day cycle
  Interventions: Drug: Tesetaxel
- Tesetaxel weekly (Experimental): Tesetaxel 15 mg/m2 orally once every 7 days for 3 consecutive weeks on Day 1, Day 8, and Day 15 in a 28-day cycle
  Interventions: Drug: Tesetaxel
- Capecitabine (Active Comparator): Capecitabine 1250 mg/m2 orally twice daily (equivalent to a total daily dose of 2500 mg/m2) on Day 1 through Day 14 in a 21-day cycle
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Tesetaxel — Tesetaxel 27 mg/m2 orally once on Day 1 of each 21-day cycle
  Arms: Tesetaxel every 3 weeks
Drug: Tesetaxel — Tesetaxel 15 mg/m2 orally once every 7 days for 3 consecutive weeks on Day 1, Day 8, and Day 15 of each 28-day cycle
  Arms: Tesetaxel weekly
Drug: Capecitabine — Capecitabine 1250 mg/m2 orally twice daily (in the morning and evening after a meal; equivalent to a total daily dose of 2500 mg/m2) on Day 1 through Day 14 of each 21-day cycle
  Other Names: Xeloda
  Arms: Capecitabine

SUMMARY:
This study is being conducted to compare the efficacy and safety of tesetaxel administered once every 3 weeks in a 21-day cycle, tesetaxel administered once weekly for 3 consecutive weeks in a 28-day cycle, and capecitabine administered twice daily for 14 consecutive days in a 21-day cycle.

ELIGIBILITY:
Key inclusion criteria:

1. Female
2. At least 18 years of age
3. Locally advanced non-resectable or metastatic breast cancer
4. HER2 negative disease
5. Measurable disease per revised RECIST, Version 1.1
6. Eastern Cooperative Oncology Group performance status 0 or 1
7. Chemotherapy naïve, OR 1 prior chemotherapy regimen in the neoadjuvant or adjuvant setting provided the patient has had a disease-free interval of ≥ 12 months after ending this chemotherapy. If the neoadjuvant or adjuvant chemotherapy included a taxane, ≥ 2 years must have passed since this treatment ended.
8. Documented disease recurrence or progression
9. Adequate bone marrow, hepatic, and renal function
10. Ability to swallow an oral solid-dosage form of medication
11. Written informed consent

Key exclusion criteria:

1. Known metastasis to the central nervous system
2. Other cancer within the preceding 5 years other than curatively treated basal or squamous cell carcinoma of the skin or carcinoma of the cervix in situ
3. Significant medical disease other than breast cancer
4. Presence of neuropathy > Grade 1 (NCI CTC)
5. History of hypersensitivity to a taxane or capecitabine, other fluoropyrimidine agents, or any of their ingredients
6. History of severe or unexpected reaction to fluoropyrimidine therapy
7. Need to continue any regularly-taken medication that is a potent inhibitor or inducer of the CYP3A pathway
8. Less than 2 weeks since use of a medication or ingestion of an agent, beverage, or food that is a potent inhibitor or inducer of the CYP3A pathway
9. Known dihydropyrimidine dehydrogenase deficiency
10. Pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-09 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Response rate | 4 months after the date of randomization of the last patient, which is estimated will occur 16 months after the first patient is randomized
  the percentage of patients with a confirmed complete or partial response, as defined in the revised Response Evaluation Criteria in Solid Tumors (revised RECIST [Version 1.1])

SECONDARY OUTCOMES:
Clinical benefit rate | 12 months after the date of randomization of the last patient, which is estimated will occur 24 months after the first patient is randomized
  the percentage of patients with a complete or partial response of any duration or stable disease lasting ≥ 6 months
Progression-free survival | 12 months after the date of randomization of the last patient, which is estimated will occur 24 months after the first patient is randomized
  the period from the date of randomization to the date when disease progression is first documented or when the patient dies within 6 weeks of the last lesion assessment
Progression-free survival rate | 6 and 12 months after patients' date of randomization
  the percentage of patients who are progression free
Adverse events | up to 30 days after patients' last dose of study medication
  the percentage of patients with adverse events classified by term and body system

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Seidman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- The West Clinic, Memphis, Tennessee, United States